CLINICAL TRIAL: NCT03638687
Title: Neuroimaging Epigenetics of Prospective Postpartum Depression Biomarkers
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00038271; R01MH104262 (NIH)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Post Partum Depression; Bipolar Disorder
Keywords: Pregnancy; Postpartum
MeSH Terms: conditions — Depression, Postpartum; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- History, Yes PPD: Participants may be asked to undergo repeated neuroimaging scans. No intervention will be administered, all participants will receive routine care during the study.
- No History, No PPD: Participants may be asked to undergo repeated neuroimaging scans. No intervention will be administered, all participants will receive routine care during the study.
- History, No PPD: Participants may be asked to undergo repeated neuroimaging scans. No intervention will be administered, all participants will receive routine care during the study.
- No History, Yes PPD: Participants may be asked to undergo repeated neuroimaging scans. No intervention will be administered, all participants will receive routine care during the study.

SUMMARY:
Through a recent cross species translational experiment, researchers have identified a set of epigenetic marks capable of predicting postpartum depression with greater than 85% accuracy. The researchers are looking to identify a group of women from both the general population and those with a history of mood disorders who are at risk for postpartum depression and obtain brain imaging data at a postpartum time period prior to the onset of depressive symptoms and compare it with those obtained during depressive episodes. The researchers will also evaluate the efficacy of postpartum depression biomarker prediction.

DETAILED DESCRIPTION:
Postpartum depression (PPD) occurs in approximately 10-18% of women from the general population, affecting ~400,000 to 800,000 women each year. PPD results in significant morbidity to both mother and child, with offspring risks including low self-esteem, low intellectual skills, child abuse, and infanticide. PPD occurs within four weeks following parturition according to Diagnostic and Statistical Manual (DSM)-IV criteria and follows a dramatic drop in the circulating levels of estradiol (E2) and progesterone (P4). While PPD risk is not predicted by serum levels of gonadal hormones in humans, numerous studies suggest that risk to PPD is mediated by hormonal sensitivity. Recently, the investigators demonstrated that women at risk to PPD demonstrate an increased sensitivity to E2 mediated DNA methylation reprogramming at hippocampally relevant genes and identified two biomarkers, Tetratricopeptide repeat protein 9B (TTC9B) and heterochromatin protein 1 binding protein 3 (HP1BP3) that appeared functionally related to modulating neuroplasticity and which were predictive of PPD with 82-96% accuracy. Given that peripherally measurable epigenetic marks in genes implicated in hormone related neuroplastic changes may underlie risk to PPD, it is logical to next investigate neuroconnectivity alterations occurring longitudinally in the postpartum population at risk for PPD. The study is divided into two waves; in wave 1, the researchers will draw a tube of blood to be used as a biomarker screening to identify those at risk for PPD and matched controls, who will be asked to enter wave 2 of the study. In wave 2, women will undergo neuroimaging at weeks 2 and 6 postpartum in hopes to gather a neural signature of PPD prior to the onset of symptoms and while experiencing the symptoms. Additionally, data on a variety of candidate moderators of depression during or after pregnancy will be collected at each visit. This includes history of premenstrual symptoms, use of oral contraceptives, use of hormonal treatments to promote pregnancy and psychiatric history during previous pregnancies and the postpartum. Several measures of mood symptoms and anxiety symptoms will be administered including: Edinburgh Postnatal Depression Rating Scale (EPDS) which measures depressive symptoms in pregnant and postpartum mothers, the Young Mania Rating Scale, which rates manic and hypomanic symptoms, and the State Trait Anxiety Inventory, Perinatal Anxiety Scale, and the Penn State Worry questionnaire which measure anxiety symptoms. The Pittsburgh Sleep Quality Index scale will be administered at every visit to assess the role of sleep in the relapse of depression in the mothers. Two scales designed to measure stress will be administered to allow examination of its potential role in Major Depressive Disorder (MDD) relapse. The Recent Life Changes Scale, which measures stressful life events, will be administered at the Screening, 3rd trimester and 6 week visits. The Perceived Stress Scale which provides a subjective rating of the stress of will be administered at every visit. The investigators will also administer measures of childhood trauma, and note demographic information, medication usage, clinical history (e.g. number of hospitalizations, medication trials, etc.) and birth outcomes. These measures will be used in future exploratory analyses of potential moderators of epigenetic changes seen during and after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 18 or older with singleton pregnancy
* with or without history of a mood disorder
* may use psychiatric or Over-the-counter (OTC) medications
* may have experienced preterm labor or delivery
* must be willing to undergo repeated MRI scans (for wave 2)

Exclusion Criteria:

* current active suicidal ideation
* medical or psychiatric instability
* active substance abuse or dependence in last 90 days
* any significant neurologic disease (wave 2)
* presence of known infection, infarction, lesion in critical memory structures of brain (wave 2)
* pace maker, aneurysm clips, artificial heart valve, ear implants, metal fragments (wave 2)
* high risk pregnancy indications i.e. preeclampsia, genetic anomalies, women with HIV, Lupus, Irritable Bowel Syndrome (IBS) (wave 2)
* implanted Intra-uterine devices (IUDs) or birth control prior to 6 weeks postpartum (wave 2)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes women 18 years or older, pregnant with a singleton pregnancy, and with or without a history of a mood disorder. Participants may take psychiatric medications, however they may not be currently suicidal, psychiatrically unstable, or be currently abusing substances.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Epigenetic Analysis | At week 33 of pregnancy
  One blood sample will be drawn in the third trimester and the epigenetic information obtained will be put into a model of prediction for postpartum depression.

SECONDARY OUTCOMES:
Brain Imaging | 4 Weeks
  An functional MRI (fMRI) of hippocampal subregions and surrounding structures at a postpartum time period prior to the onset of depressive symptoms (2 weeks postpartum) and compared with those obtained during depressive episodes (6 weeks postpartum) to assess differences in functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary A Kaminsky, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins East Baltimore Medical Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Hara MW. Postpartum depression: what we know. J Clin Psychol. 2009 Dec;65(12):1258-69. doi: 10.1002/jclp.20644. PMID 19827112
- [Background] Soufia M, Aoun J, Gorsane MA, Krebs MO. [SSRIs and pregnancy: a review of the literature]. Encephale. 2010 Dec;36(6):513-6. doi: 10.1016/j.encep.2010.02.003. Epub 2010 Apr 3. French. PMID 21130237
- [Background] Field T. Prenatal depression effects on early development: a review. Infant Behav Dev. 2011 Feb;34(1):1-14. doi: 10.1016/j.infbeh.2010.09.008. PMID 20970195
- [Background] Breese McCoy SJ. Postpartum depression: an essential overview for the practitioner. South Med J. 2011 Feb;104(2):128-32. doi: 10.1097/SMJ.0b013e318200c221. PMID 21206417
- [Background] Cuijpers P, Brannmark JG, van Straten A. Psychological treatment of postpartum depression: a meta-analysis. J Clin Psychol. 2008 Jan;64(1):103-18. doi: 10.1002/jclp.20432. PMID 18161036
- [Background] Hirst KP, Moutier CY. Postpartum major depression. Am Fam Physician. 2010 Oct 15;82(8):926-33. PMID 20949886
- [Background] Marcus SM. Depression during pregnancy: rates, risks and consequences--Motherisk Update 2008. Can J Clin Pharmacol. 2009 Winter;16(1):e15-22. Epub 2009 Jan 22. PMID 19164843
- [Background] Studd JW. A guide to the treatment of depression in women by estrogens. Climacteric. 2011 Dec;14(6):637-42. doi: 10.3109/13697137.2011.609285. Epub 2011 Aug 31. PMID 21878053
- [Background] Bloch M, Schmidt PJ, Danaceau M, Murphy J, Nieman L, Rubinow DR. Effects of gonadal steroids in women with a history of postpartum depression. Am J Psychiatry. 2000 Jun;157(6):924-30. doi: 10.1176/appi.ajp.157.6.924. PMID 10831472
- [Background] Bloch M, Rubinow DR, Schmidt PJ, Lotsikas A, Chrousos GP, Cizza G. Cortisol response to ovine corticotropin-releasing hormone in a model of pregnancy and parturition in euthymic women with and without a history of postpartum depression. J Clin Endocrinol Metab. 2005 Feb;90(2):695-9. doi: 10.1210/jc.2004-1388. Epub 2004 Nov 16. PMID 15546899
- [Background] Guintivano J, Arad M, Gould TD, Payne JL, Kaminsky ZA. Antenatal prediction of postpartum depression with blood DNA methylation biomarkers. Mol Psychiatry. 2014 May;19(5):560-7. doi: 10.1038/mp.2013.62. Epub 2013 May 21. PMID 23689534
- [Background] Kimmel M, Kaminsky Z, Payne JL. Biomarker or pathophysiology? The role of DNA methylation in postpartum depression. Epigenomics. 2013;5(5):473-5. doi: 10.2217/epi.13.51. No abstract available. PMID 24059792
- [Background] Walf AA, Koonce CJ, Frye CA. Estradiol or diarylpropionitrile decrease anxiety-like behavior of wildtype, but not estrogen receptor beta knockout, mice. Behav Neurosci. 2008 Oct;122(5):974-81. doi: 10.1037/a0012749. PMID 18823154
- [Background] Osterlund MK, Witt MR, Gustafsson JA. Estrogen action in mood and neurodegenerative disorders: estrogenic compounds with selective properties-the next generation of therapeutics. Endocrine. 2005 Dec;28(3):235-42. doi: 10.1385/ENDO:28:3:235. PMID 16388113
- [Background] Lund TD, Rovis T, Chung WC, Handa RJ. Novel actions of estrogen receptor-beta on anxiety-related behaviors. Endocrinology. 2005 Feb;146(2):797-807. doi: 10.1210/en.2004-1158. Epub 2004 Oct 28. PMID 15514081
- [Background] Walf AA, Rhodes ME, Frye CA. Antidepressant effects of ERbeta-selective estrogen receptor modulators in the forced swim test. Pharmacol Biochem Behav. 2004 Jul;78(3):523-9. doi: 10.1016/j.pbb.2004.03.023. PMID 15251261
- [Background] Walf AA, Frye CA. ERbeta-selective estrogen receptor modulators produce antianxiety behavior when administered systemically to ovariectomized rats. Neuropsychopharmacology. 2005 Sep;30(9):1598-609. doi: 10.1038/sj.npp.1300713. PMID 15798780
- [Background] Tanaka M, Sokabe M. Bidirectional modulatory effect of 17beta-estradiol on NMDA receptors via ERalpha and ERbeta in the dentate gyrus of juvenile male rats. Neuropharmacology. 2013 Dec;75:262-73. doi: 10.1016/j.neuropharm.2013.07.029. Epub 2013 Aug 14. PMID 23954493
- [Background] Van Kempen TA, Kahlid S, Gonzalez AD, Spencer-Segal JL, Tsuda MC, Ogawa S, McEwen BS, Waters EM, Milner TA. Sex and estrogen receptor expression influence opioid peptide levels in the mouse hippocampal mossy fiber pathway. Neurosci Lett. 2013 Sep 27;552:66-70. doi: 10.1016/j.neulet.2013.07.048. Epub 2013 Aug 7. PMID 23933204
- [Background] MacLusky NJ, Luine VN, Hajszan T, Leranth C. The 17alpha and 17beta isomers of estradiol both induce rapid spine synapse formation in the CA1 hippocampal subfield of ovariectomized female rats. Endocrinology. 2005 Jan;146(1):287-93. doi: 10.1210/en.2004-0730. Epub 2004 Oct 14. PMID 15486220
- [Background] ter Horst GJ. Estrogen in the limbic system. Vitam Horm. 2010;82:319-38. doi: 10.1016/S0083-6729(10)82017-5. PMID 20472146
- [Background] Fester L, Labitzke J, Hinz R, Behem C, Horling K, Bernhard T, Bader MI, Vollmer G, Rune GM. Estradiol responsiveness of synaptopodin in hippocampal neurons is mediated by estrogen receptor beta. J Steroid Biochem Mol Biol. 2013 Nov;138:455-61. doi: 10.1016/j.jsbmb.2013.09.004. Epub 2013 Sep 25. PMID 24076016
- [Background] Suda S, Segi-Nishida E, Newton SS, Duman RS. A postpartum model in rat: behavioral and gene expression changes induced by ovarian steroid deprivation. Biol Psychiatry. 2008 Aug 15;64(4):311-9. doi: 10.1016/j.biopsych.2008.03.029. Epub 2008 May 8. PMID 18471802
- [Background] Green AD, Galea LA. Adult hippocampal cell proliferation is suppressed with estrogen withdrawal after a hormone-simulated pregnancy. Horm Behav. 2008 Jun;54(1):203-11. doi: 10.1016/j.yhbeh.2008.02.023. Epub 2008 Mar 12. PMID 18423635
- [Background] Bennett MR. The prefrontal-limbic network in depression: Modulation by hypothalamus, basal ganglia and midbrain. Prog Neurobiol. 2011 Apr;93(4):468-87. doi: 10.1016/j.pneurobio.2011.01.006. Epub 2011 Feb 22. PMID 21349315
- [Background] Taylor SF, Liberzon I. Neural correlates of emotion regulation in psychopathology. Trends Cogn Sci. 2007 Oct;11(10):413-8. doi: 10.1016/j.tics.2007.08.006. PMID 17928261
- [Background] Silverman ME, Loudon H, Safier M, Protopopescu X, Leiter G, Liu X, Goldstein M. Neural dysfunction in postpartum depression: an fMRI pilot study. CNS Spectr. 2007 Nov;12(11):853-62. doi: 10.1017/s1092852900015595. PMID 17984858
- [Background] Moses-Kolko EL, Perlman SB, Wisner KL, James J, Saul AT, Phillips ML. Abnormally reduced dorsomedial prefrontal cortical activity and effective connectivity with amygdala in response to negative emotional faces in postpartum depression. Am J Psychiatry. 2010 Nov;167(11):1373-80. doi: 10.1176/appi.ajp.2010.09081235. Epub 2010 Sep 15. PMID 20843875
- [Background] Leibenluft E, Yonkers KA. The ties that bind: maternal-infant interactions and the neural circuitry of postpartum depression. Am J Psychiatry. 2010 Nov;167(11):1294-6. doi: 10.1176/appi.ajp.2010.10081159. No abstract available. PMID 21041250
- [Background] Barrett J, Wonch KE, Gonzalez A, Ali N, Steiner M, Hall GB, Fleming AS. Maternal affect and quality of parenting experiences are related to amygdala response to infant faces. Soc Neurosci. 2012;7(3):252-68. doi: 10.1080/17470919.2011.609907. Epub 2011 Sep 26. PMID 21943083
- [Background] Laurent HK, Ablow JC. A face a mother could love: depression-related maternal neural responses to infant emotion faces. Soc Neurosci. 2013;8(3):228-39. doi: 10.1080/17470919.2012.762039. Epub 2013 Jan 21. PMID 23330663
- [Background] Deligiannidis KM, Sikoglu EM, Shaffer SA, Frederick B, Svenson AE, Kopoyan A, Kosma CA, Rothschild AJ, Moore CM. GABAergic neuroactive steroids and resting-state functional connectivity in postpartum depression: a preliminary study. J Psychiatr Res. 2013 Jun;47(6):816-28. doi: 10.1016/j.jpsychires.2013.02.010. Epub 2013 Mar 15. PMID 23499388
- [Background] Bannbers E, Gingnell M, Engman J, Morell A, Sylven S, Skalkidou A, Kask K, Backstrom T, Wikstrom J, Poromaa IS. Prefrontal activity during response inhibition decreases over time in the postpartum period. Behav Brain Res. 2013 Mar 15;241:132-8. doi: 10.1016/j.bbr.2012.12.003. Epub 2012 Dec 10. PMID 23238040
- [Background] Amin Z, Epperson CN, Constable RT, Canli T. Effects of estrogen variation on neural correlates of emotional response inhibition. Neuroimage. 2006 Aug 1;32(1):457-64. doi: 10.1016/j.neuroimage.2006.03.013. Epub 2006 Apr 27. PMID 16644236
- [Background] Guy, W., Clinical global impression. ECDEU Assessment Manual for Psychopharmacology, Revised. 1976, Rockville, MD: National Institute of Mental Health.
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Lee KA. Self-reported sleep disturbances in employed women. Sleep. 1992 Dec;15(6):493-8. doi: 10.1093/sleep/15.6.493. PMID 1475563
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Costa PT Jr, McCrae RR. Domains and facets: hierarchical personality assessment using the revised NEO personality inventory. J Pers Assess. 1995 Feb;64(1):21-50. doi: 10.1207/s15327752jpa6401_2. PMID 16367732
- [Background] Magiakou MA, Mastorakos G, Rabin D, Dubbert B, Gold PW, Chrousos GP. Hypothalamic corticotropin-releasing hormone suppression during the postpartum period: implications for the increase in psychiatric manifestations at this time. J Clin Endocrinol Metab. 1996 May;81(5):1912-7. doi: 10.1210/jcem.81.5.8626857.
- [Background] Stuebe AM, Grewen K, Pedersen CA, Propper C, Meltzer-Brody S. Failed lactation and perinatal depression: common problems with shared neuroendocrine mechanisms? J Womens Health (Larchmt). 2012 Mar;21(3):264-72. doi: 10.1089/jwh.2011.3083. Epub 2011 Dec 28. PMID 22204416
- [Background] Bunevicius R, Kusminskas L, Mickuviene N, Bunevicius A, Pedersen CA, Pop VJ. Depressive disorder and thyroid axis functioning during pregnancy. World J Biol Psychiatry. 2009;10(4):324-9. doi: 10.3109/15622970903144038. PMID 19921974
- [Background] Pedersen CA, Johnson JL, Silva S, Bunevicius R, Meltzer-Brody S, Hamer RM, Leserman J. Antenatal thyroid correlates of postpartum depression. Psychoneuroendocrinology. 2007 Apr;32(3):235-45. doi: 10.1016/j.psyneuen.2006.12.010. Epub 2007 Mar 7. PMID 17346901
- [Background] Skrundz M, Bolten M, Nast I, Hellhammer DH, Meinlschmidt G. Plasma oxytocin concentration during pregnancy is associated with development of postpartum depression. Neuropsychopharmacology. 2011 Aug;36(9):1886-93. doi: 10.1038/npp.2011.74. Epub 2011 May 11. PMID 21562482
- [Background] Andreen L, Nyberg S, Turkmen S, van Wingen G, Fernandez G, Backstrom T. Sex steroid induced negative mood may be explained by the paradoxical effect mediated by GABAA modulators. Psychoneuroendocrinology. 2009 Sep;34(8):1121-32. doi: 10.1016/j.psyneuen.2009.02.003. Epub 2009 Mar 9. PMID 19272715
- [Background] Backstrom T, Haage D, Lofgren M, Johansson IM, Stromberg J, Nyberg S, Andreen L, Ossewaarde L, van Wingen GA, Turkmen S, Bengtsson SK. Paradoxical effects of GABA-A modulators may explain sex steroid induced negative mood symptoms in some persons. Neuroscience. 2011 Sep 15;191:46-54. doi: 10.1016/j.neuroscience.2011.03.061. Epub 2011 May 13. PMID 21600269
- [Background] Yim IS, Glynn LM, Schetter CD, Hobel CJ, Chicz-Demet A, Sandman CA. Prenatal beta-endorphin as an early predictor of postpartum depressive symptoms in euthymic women. J Affect Disord. 2010 Sep;125(1-3):128-33. doi: 10.1016/j.jad.2009.12.009. Epub 2010 Jan 3. PMID 20051292
- [Background] Kahn I, Andrews-Hanna JR, Vincent JL, Snyder AZ, Buckner RL. Distinct cortical anatomy linked to subregions of the medial temporal lobe revealed by intrinsic functional connectivity. J Neurophysiol. 2008 Jul;100(1):129-39. doi: 10.1152/jn.00077.2008. Epub 2008 Apr 2. PMID 18385483
- [Background] Bakker A, Krauss GL, Albert MS, Speck CL, Jones LR, Stark CE, Yassa MA, Bassett SS, Shelton AL, Gallagher M. Reduction of hippocampal hyperactivity improves cognition in amnestic mild cognitive impairment. Neuron. 2012 May 10;74(3):467-74. doi: 10.1016/j.neuron.2012.03.023. PMID 22578498
- [Background] Yassa MA, Stark SM, Bakker A, Albert MS, Gallagher M, Stark CE. High-resolution structural and functional MRI of hippocampal CA3 and dentate gyrus in patients with amnestic Mild Cognitive Impairment. Neuroimage. 2010 Jul 1;51(3):1242-52. doi: 10.1016/j.neuroimage.2010.03.040. Epub 2010 Mar 23. PMID 20338246
- [Background] Lacy JW, Yassa MA, Stark SM, Muftuler LT, Stark CE. Distinct pattern separation related transfer functions in human CA3/dentate and CA1 revealed using high-resolution fMRI and variable mnemonic similarity. Learn Mem. 2010 Dec 16;18(1):15-8. doi: 10.1101/lm.1971111. Print 2011 Jan. PMID 21164173
- [Background] Avants BB, Yushkevich P, Pluta J, Minkoff D, Korczykowski M, Detre J, Gee JC. The optimal template effect in hippocampus studies of diseased populations. Neuroimage. 2010 Feb 1;49(3):2457-66. doi: 10.1016/j.neuroimage.2009.09.062. Epub 2009 Oct 8. PMID 19818860
- [Background] Klein A, Andersson J, Ardekani BA, Ashburner J, Avants B, Chiang MC, Christensen GE, Collins DL, Gee J, Hellier P, Song JH, Jenkinson M, Lepage C, Rueckert D, Thompson P, Vercauteren T, Woods RP, Mann JJ, Parsey RV. Evaluation of 14 nonlinear deformation algorithms applied to human brain MRI registration. Neuroimage. 2009 Jul 1;46(3):786-802. doi: 10.1016/j.neuroimage.2008.12.037. Epub 2009 Jan 13. PMID 19195496
- [Background] Bakker A, Kirwan CB, Miller M, Stark CE. Pattern separation in the human hippocampal CA3 and dentate gyrus. Science. 2008 Mar 21;319(5870):1640-2. doi: 10.1126/science.1152882. PMID 18356518
- [Background] Pinette MG, Wax JR. The management of depression during pregnancy: a report from the American Psychiatric Association and the American College of Obstetricians and Gynecologists. Obstet Gynecol. 2010 Jan;115(1):188-189. doi: 10.1097/AOG.0b013e3181c8b21d. No abstract available. PMID 20027064